CLINICAL TRIAL: NCT06335186
Title: Predictive and Prognostic Significance of Age,Blood Tests,Comorbidities(ABC) Score,Cologne Watch(C-watch)Score and Rockall Score for Risk of Variceal Re-bleeding Among Cirrhotic Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Sayed Ahmed, Resident in Tropical Medicine and gastroenterology department, Sohag University
Other Study IDs: Soh-Med-24-03-04MS
Record Dates: First submitted 2024-03-20; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Upper Gastrointestinal Variceal Bleeding in Cirrhotic Patients
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: upper endoscopy — to detect esophageal or gastric varices

SUMMARY:
Introduction

Portal hypertension is a common complication of liver cirrhosis and is often underestimated in clinical diagnosis. The incidence of portal hypertension is approximately 20% to 98% in patients with cirrhosis (Wu et al., 2022). It is the major driver in the transition from the compensated to the 'decompensated' stage of cirrhosis, defined by the presence of clinical complications, including ascites, spontaneous bacterial peritonitis, hepatorenal syndrome, and hepatic encephalopathy (Berzigotti., 2017).

Acute variceal bleeding is one of the most lifethreatening complications of liver cirrhosis. Twenty two percent to sixty one percent of cirrhotic patients receiving primary prophylaxis will develop first variceal bleeding during the first two years of follow up. Furthermore, variceal bleeding is associated with high risk of rebleeding and mortality (Tantai et al., 2019).

Patients with cirrhosis, although much progress has been made in diagnosis and treatment using vasoactive drugs, preventive antibiotics, early endoscopy and interventional radiology, the 6-week mortality rate remains high, ranging from 10 to 20%, mainly due to failure to control bleeding in the first days. Therefore, the prognostic method of patients with acute variceal bleeding is to determine the risk of rebleeding and resistance to standard treatment (accounting for 20-30%) and mortality rate in order to be able to adopt more aggressive treatment measures. The prognosis is very important but also difficult, not only because of the bleeding status but also depending on the severity of the underlying cirrhosis (Huy et al., 2023).

Many risk factors are known to influence the outcome in Upper Gastrointestinal Bleeding (UGIB) setting: Age, comorbidities, presence of shock, endoscopic diagnosis, haemoglobin values at the time of bleeding, stigmata of recent haemorhage and need for blood transfusion have all been described as significant risk factors for rebleeding and death (Monteiro S et al., 2016).

Many risk assessment score systems, including pre-endoscopy and post-endoscopy evaluations, have been developed to predict outcomes such as the need for hospital-based intervention, endoscopic therapy, and admission to an intensive care unit (ICU), rebleeding, and mortality. Some studies showed that these scoring systems distinguish low-risk patients who can potentially be managed as outpatients, allowing more efficient use of resources. Other studies suggested that these score systems distinguish higher-risk patients who might require emergency endoscopy or management in an intensive care unit (Li et al., 2022).

In 1993, the Rockall Scoring system was introduced to predict the mortality after UGIB and was validated for its use to identify the patients at high risk for re-bleed and mortality. Complete Rockall scoring system is based on an initial clinical score at the time of admission which consist of age (score 0-2), presence of shock (0-2), co-morbidities (score 0-3) and post endoscopic diagnosis (score 0-2) with stigmata of recent hemorrhages (score 0-2). Both clinical and post endoscopic scores added together gives a complete Rockall score with maximum score being 11 (Dewan et al., 2018).

In 2020, Laursen S.B. and colleagues conducted a multicenter international study and developed a new prognostic scoring system for UGIB called the ABC score. This scoring system is based on three criteria: age, blood test results, and comorbidities. The score ranges from 0 to 18 points, categorizing the risk into low (≤3 points), moderate (4-7 points), and high (≥8 points) levels. The 30-day mortality rates for high-risk UGIB patients in these three risk groups were 1%, 7%, and 25%, respectively ( Ky et al., 2023)

The new Cologne Watch (C-Watch) score was designed as a pre-endoscopic score for acute variceal and non-variceal UGIB and incorporates laboratory values only (c-reactive protein, white blood cell count, alanine-aminotransferase, thrombocytes, creatinine, and hemoglobin) with a minimum point value of 0 and a maximum point value of 8. Within the validation set, it predicted a composite endpoint consisting of recurrent bleeding, need for intervention (interventional radiology, surgery), or death within 30 days with an area under the receiver-operating characteristics curve (AUROC) of 0. About 38.7% of patients were within the high-risk group, i.e., ≥2 points, reached the composite endpoint, whereas no patient classified as low risk (≤1 point) (Allo et al., 2022).

DETAILED DESCRIPTION:
Patients and methods

-Place of the study

Tropical Medicine and Gastroenterology Department of Sohag University Hospital.

-Type of the study

Prospective cohort study.

-Study period

Duration of study will be one year after protocol acceptance.

-Patients

This study will include 100 cirrhotic Patients presenting with upper gastrointestinal variceal bleeding.

-Inclusion criteria

Patients who met the following inclusion criteria were enrolled:

1-History of chronic liver disease. 2-Impaired liver function. 3-Portal hypertension syndrome (indicated by esophageal varices and/or variceal dilation).

4-Diagnostic imaging confirming liver cirrhosis on ultrasound who admitted to the hospital with symptoms of hematemesis and/or melena underwent clinical and laboratory examinations and an upper gastrointestinal endoscopy and were diagnosed with UGIB due to ruptured esophageal (ESOVs) and/or gastric varices (GASVs).

* Exclusion criteria

  1. UGIB caused by other cases such as Mallory-Weiss syndrome and esophageal or gastrointestinal ulcers.
  2. UGIB due to ruptured veins in conditions other than increased portal pressure like portal hypertension syndrome unrelated to cirrhosis.
  3. Patients with portal vein thrombosis.
  4. Patients used anticoagulant.
* Methods of the study

All participants will be subjected to:

* Complete history taking.
* Clinical examination:

  1. Vital signs (pulse 60-100, blood pressure 90/60-120/80 and temperature 36.5-37.3).
  2. Complete general and local examination.
* Laboratory investigation:

  1. Complete blood count (Hemoglobin (Hb), white blood cells (WBC) and platelet).
  2. Liver function test as alanine transaminase (ALT), aspartate transaminase (AST), Albumin, total bilirubin, Prothrombin time (PT), Prothrombin concentration (PC), International normalized ratio (INR) and child pugh score).
  3. Serum creatinine,urea and C-reactive protein (CRP).
  4. Ascitic fluid study for patients with ascites.
* Assessment of risk and predicting outcomes by:

  1. ABC score.
  2. C-watch score.
  3. Rockall score.

     * Radiological investigation

Abdominal ultrasound with comment on:

* Liver size, echopattern, surface and focal lesion.
* Portal vein diameter, patency and presence of collaterals.
* Spleen size, echopattern and splenic vein diameter.
* Presence of ascites or not.

  * Intervention:

Upper endoscopy with comment on:

* Size of varices, extension of varices and stigmata of recent bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the following inclusion criteria were enrolled:

  1. History of chronic liver disease.
  2. Impaired liver function.
  3. Portal hypertension syndrome (indicated by esophageal varices and/or variceal dilation).
  4. Diagnostic imaging confirming liver cirrhosis on ultrasound who admitted to the hospital with symptoms of hematemesis and/or melena underwent clinical and laboratory examinations and an upper gastrointestinal endoscopy and were diagnosed with UGIB due to ruptured esophageal (ESOVs) and/or gastric varices (GASVs).

     Exclusion Criteria:
* Exclusion criteria

  1. UGIB caused by other cases such as Mallory-Weiss syndrome and esophageal or gastrointestinal ulcers.
  2. UGIB due to ruptured veins in conditions other than increased portal pressure like portal hypertension syndrome unrelated to cirrhosis.
  3. Patients with portal vein thrombosis.
  4. Patients used anticoagulan

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who met the following inclusion criteria were enrolled:
  1. History of chronic liver disease.
  2. Impaired liver function.
  3. Portal hypertension syndrome (indicated by esophageal varices and/or variceal dilation).
  4. Diagnostic imaging confirming liver cirrhosis on ultrasound who admitted to the hospital with symptoms of hematemesis and/or melena underwent clinical and laboratory examinations and an upper gastrointestinal endoscopy and were diagnosed with UGIB due to ruptured esophageal (ESOVs) and/or gastric varices (GASVs).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
ABC score. | 1 year
  To predict risk of variceal rebleeding in cirrhotic patient.
Rockall score | 1 year
  To predict outcome of variceal bleeding in cirrhotic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berzigotti A. Advances and challenges in cirrhosis and portal hypertension. BMC Med. 2017 Nov 10;15(1):200. doi: 10.1186/s12916-017-0966-6. PMID 29121925
- [Background] Ky TD, Trang NTH, Binh MT. Predictive Significance of the ABC Score for Early Re-Hemorrhage and In-Hospital Mortality in High-Risk Variceal Bleeding among Cirrhotic Patients. Diagnostics (Basel). 2023 Nov 29;13(23):3570. doi: 10.3390/diagnostics13233570. PMID 38066811
- [Background] Monteiro S, Goncalves TC, Magalhaes J, Cotter J. Upper gastrointestinal bleeding risk scores: Who, when and why? World J Gastrointest Pathophysiol. 2016 Feb 15;7(1):86-96. doi: 10.4291/wjgp.v7.i1.86. PMID 26909231
- [Background] Tantai XX, Liu N, Yang LB, Wei ZC, Xiao CL, Song YH, Wang JH. Prognostic value of risk scoring systems for cirrhotic patients with variceal bleeding. World J Gastroenterol. 2019 Dec 7;25(45):6668-6680. doi: 10.3748/wjg.v25.i45.6668. PMID 31832005